CLINICAL TRIAL: NCT07323836
Title: Effect Of Mckenzie Exercises On Postural Stability In Mechanical Back Pain Patients With Prolonged Sitting Posture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Samir Gomaa Shahat, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/006115
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: MECHANICAL BACK PAIN
Keywords: MCKENZIE EXERCISES; POSTURAL STABILITY; MECHANICAL BACK PAIN; PROLONGED SITTING POSTURE

STUDY DESIGN:
Intervention Model Description: Mackenzie exercises vs traditional physiotherapy program
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mckenzie exercise (Experimental): this group will receive traditional physiotherapy program plus, Exercise 1 lying prone the patient adopts the prone lying position with the arms alongside the trunk and the head turns to one side. Exercise 2 lying prone in extension places the elbows under the shoulders and raises the top half of his body so that he comes to lean on elbows and forearms while pelvis and thighs remain on the couch. .Exercise 3 extension in lying the patient, already lying prone, places the hands (palms down) near the shoulders as for the traditional press-up exercise. and the exercise is repeated about ten times.Exercise 4 extension in standing the patient stands with the feet well apart and place the hands (fingers pointing backwards) in the small of the back across the belt line. He leans backwards as far as possible, using the hands as a fulcrum, and then returns to neutral standing. The exercise is repeated about ten times.
  Interventions: Other: mckenzie exercises
- traditional physiotherapy program (Active Comparator): traditional physiotherapy program is composed of 1-TENS:pulse frequencies>250 pulses per second (pps), pulse durations>500 microseconds (µs) and peak-to-peak amplitudes>60 milliamperes (mA), pulse frequency from 0.7 to 108 Hz and a pulse width of 100 μs. Intensity level was instructed to be as high as tolerable.2-Hot pack: heated wrap applied for eight hours, or an electric blanket applied for 25 minutes, and at (104 -113) degree Fahrenheit.3-Ultrasound : 1 or 3 MHz and at amplitude densities between 0.1 W/cm² and 3 W/cm².pulsed.4-strengthening exercises: The exercise program includes a warm-up session (awareness of the back, pelvic tilt, whole-body movement in standing), back extensors, posterior buttocks, abdominals, lateral buttocks, leg muscles, as well as exercises for flexibility. Exercise will be at 60-70% of one repetition maximum (RM), held for 30 s and repeated 2-4 time.
  Interventions: Other: mckenzie exercises

INTERVENTIONS:
Other: mckenzie exercises — they will receive traditional physiotherapy program (transcutaneous electrical nerve stimulation, heat therapy, ultrasound and strengthening exercises) plus Mckenzie
  Other Names: traditional physiotherapy program

SUMMARY:
Postural stability is a complex sensorimotor process that depends on the integration of visual, vestibular, and somatosensory inputs, and its impairment increases the risk of falls and negatively affects quality of life.

Prolonged sitting and low physical activity negatively influence postural stability, whereas regular physical activity has a positive chronic effect, despite some exercises causing temporary instability due to fatigue.

Breaking up sitting time with light walking or active workstations may improve postural stability, and this study aims to evaluate the effects of McKenzie back extension exercises on postural stability, pain, and quality of life in individuals with mechanical back pain.

DETAILED DESCRIPTION:
Maintaining postural stability is a sensorimotor process that involves the functional integration of sensory afferent information from the visual, vestibular, and somatosensory systems, central processing of this sensory input, and the selection of appropriate motor responses. Impaired postural stability is a major risk factor for falls and can negatively influence social interaction and mental health, particularly in older adults.

Impairment in lumbar repositioning sense, referred to as lumbar repositioning error (LRPE), may lead to poor postural habits, loss of neutral spine alignment, and reduced mechanical efficiency of the trunk muscles. Proprioception is considered the most critical sensory system for maintaining postural stability, especially under normal fixed-surface conditions. Low levels of physical activity have also been associated with an increased risk of falls, even in younger adults.

Because physical activity influences all levels of the sensorimotor system, postural stability represents an important health variable for understanding the effects of prolonged sitting. While even low-intensity physical activity may cause a short-term reduction in postural stability, regular physical activity has a positive long-term effect. Exercise impacts sensory input, central processing, and motor output, although fatigue from endurance activities can acutely reduce postural stability.

Prolonged sitting is common in modern desk-based occupations, and lack of time is a major barrier to interrupting sedentary behavior. Active workstations, such as standing desks and treadmill desks, offer a practical way to integrate physical activity into the workday and have demonstrated benefits for body composition, metabolic health, quality of life, work performance, and cognition.

Breaking up prolonged sitting with light-intensity treadmill desk walking has been shown to improve postural stability by reducing mediolateral and anteroposterior center of pressure sway. These findings suggest that treadmill desks or regular walking breaks may provide additional neuromuscular benefits beyond general health improvements. In contrast, interrupting prolonged sitting with short bouts of bodyweight resistance exercises may produce some physiological benefits but can negatively affect postural stability.

Therefore, this study aims to evaluate the effects of McKenzie back extension exercises on postural stability, pain, and quality of life in individuals with mechanical low back pain who engage in prolonged sitting, such as office workers, computer engineers, and college students, with potential implications for both physical well-being and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* • patients with mechanical Low back pain aged 18 - 35 years.

  * patients who spend at least 6 hours daily sitting (in office, at home, or screen time).
  * patients who feel some sort of discomfort and pain after prolonged sitting.
  * Patients with flat lumbar curves.
  * patients have not received any physical therapy or medications in the last six months.
  * Subjects with normal body mass index (BMI) from 18.5-24.9 kg/m2

Exclusion Criteria:

* • patients with known neurological disorders or balance disorders.

  * patients who engage in regular physical activity exceeding 150 minutes per week (as this could influence balance).
  * patients who do not sit for prolonged periods of time habitually.
  * Major structural spinal deformities (scoliosis or stenosis) inflammatory diseases
  * Sequestered hernias.
  * History of spinal surgery.
  * Lower limb and pelvis deformities e.g. Leg length discrepancy
  * patients have Severe medical or psychiatric disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
postural stability | up to 6 weeks
  postural stability will be measured by Biodex Balance System SD
pain intensity | up to 6 weeks
  pain intensity will be measured by VAS. A horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state.

SECONDARY OUTCOMES:
short form 36 health survey questionnaire (SF-36) | up to 6 weeks
  short form health survey with only 36 questions it yields an 8-scale profile of functional health and well-being scores
Arabic sedentary behaviors questionnaire (ASBQ) | up to 6 weeks
  ASBQ included a total of 16 questions providing overall as well as specific SB estimates during a variety of sedentary activities while covering leisure-time activities, work, transport, household seated activities, reading, chatting, and listening to religious verses or music.
lumbar lordotic curve by using Kinovea software program | up to 6 weeks
  The subjects stand sideways and barefoot on the back of the calibration plane with shoulders and elbows at 90°-flexion, The angle of the intersection of the lines was measured by Kinovea and decreases from 180°. The calculated angle was reported as the lordosis angle

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamèd Samir, Giza, Egypt